CLINICAL TRIAL: NCT04944199
Title: Impact of Increased Physical Activity in Young Adult Asthmatic Patients on Patient Perception of Pulmonary Health and Exercise
Brief Title: Asthma Control: Increased Physical Activity in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Jason Woloski, Clinical Assistant Professor Family Medicine, Geisinger Commonwealth School of Medicine; Assistant Program Director, Geisinger Kistler Family Medicine Residency; Principal Investigator, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-0434
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Asthma in Young Adults
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention)
- Intervention Group (Active Comparator)
  Interventions: Other: Physical Activity

INTERVENTIONS:
Other: Physical Activity — Intervention group participants will be enrolled in a standardized step-based program to gradually increase their physical activity. Daily steps will be measured via a pedometer application on a smartphone or wearable device, with a gradual increase in the goal on a weekly basis, with a target intervention of around 4-6 weeks in total. The first week's step count will be used to calculate a baseline step count for the week. At the start of each week, the participants will be asked to increase their daily step counts by 1,000.
  Arms: Intervention Group

SUMMARY:
Investigators want to study to see if patients who participate in a physical activity intervention involving increasing daily step counts will have better mini asthma quality of life questionnaire (Mini AQLQ) scores at the end of the study period compared to patients that are in the control group and do not increase daily step counts. Participants will be randomized into the two groups.

DETAILED DESCRIPTION:
The Control group (usual care group) of 75 patients will not participate in the intervention but will take an asthma control survey at baseline (point of enrollment into the study) and about 4-6 weeks after.

The Intervention group of 75 patients who will participate in the intervention of step counts and take an asthma control survey at baseline (point of enrollment into the study) and about 4-6 weeks after.

ELIGIBILITY:
Inclusion Criteria:

* Patients within the Geisinger South Wilkes-Barre Primary Care clinic with a diagnosis of mild to moderate asthma

Exclusion Criteria:

* Patients with any medical history which would prohibit their ability to participate in increased exercise, and/or patients that are diagnosed or associated with severe asthma

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Change in the Mini Asthma Quality of Life Questionnaire Score as a result of increased physical activity. | 6 weeks
  Any improvement in the score will be considered an improvement, since other than physical activity changes via step counts no other pharmacologic or lifestyle intervention will be made. Results will be compared to a control group who complete the survey without any intervention at two dates separated in time. Improvement in asthma symptoms can improve quality of life for participants. As noted by developers of the questionnaire being used in this study, "the Asthma Quality of Life Questionnaire has been developed to measure the functional (physical, emotional, occupational and social) problems that are most troublesome to adults with asthma … the impact that asthma has on a patient's quality of life cannot be inferred from the clinical indices." Descriptive statistics including means, standard deviations, medians, and interquartile ranges for continuous variables and frequency counts and percentages for categorical variables will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Woloski, MD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger South Wilkes-Barre Primary Care Clinic, Wilkes-Barre, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No